CLINICAL TRIAL: NCT01855724
Title: Phase II Single-arm Study of First Line Treatment With Gemcitabine and Pazopanib in Patients With Inoperable Locally Advanced or Metastatic Biliary Tree Cancer (Cholangiocarcinoma or Gallbladder Carcinoma)
Brief Title: Clinical Trial to Investigate the Efficacy of Treatment With Gemcitabine/Pazopanib in Patients With Biliary Tree Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE 37/12; 2012-001705-24 (EudraCT Number)
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2017-09

CONDITIONS: Cholangiocarcinoma; Gallbladder Carcinoma; Biliary Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Gallbladder Neoplasms | interventions — Gemcitabine; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine-Pazopanib (Experimental): Gemcitabine 1000 mg/m2 administered intravenously on days 1 and 8 and Pazopanib 800 mg administered per os on days 1 to 21 every 21 days.
  Treatment with gemcitabine/pazopanib combination will continue until disease progression, appearance of significant toxicity, completion of 8 cycles or informed consent withdrawal.
  Upon completion of 8 treatment cycles with the combination, and in the absence of disease progression, administration of pazopanib monotherapy as maintenance treatment will be continued until disease progression, appearance of significant toxicity or informed consent withdrawal.
  Interventions: Drug: Gemcitabine-Pazopanib

INTERVENTIONS:
Drug: Gemcitabine-Pazopanib
  Other Names: Gemzar; Votrient

SUMMARY:
The purpose of this study is to determine whether gemcitabine and pazopanib are effective in the treatment of inoperable, locally advanced or metastatic biliary tree cancer (cholangiocarcinoma or gallbladder carcinoma).

DETAILED DESCRIPTION:
This is an open label, uncontrolled, multicenter, phase II study to evaluate the efficacy and safety of Gemcitabine/Pazopanib combination as 1st line treatment in patients with unresectable, locally advanced or metastatic biliary tree adenocarcinoma. A total of 46 patients will be included in the study. The patients will receive open label Gemcitabine 1000 mg/m2 intravenously on days 1 and 8 and Pazopanib 800 mg per os on days 1 to 21 every 21 days. Treatment with gemcitabine/pazopanib combination will continue until disease progression, appearance of significant toxicity, completion of 8 cycles or informed consent withdrawal. Upon completion of 8 treatment cycles with the combination, and in the absence of disease progression, administration of pazopanib monotherapy as maintenance treatment will be continued until disease progression, appearance of significant toxicity or informed consent withdrawal.

Imaging assessments will be performed every 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments,and must be willing to comply with treatment and follow up.
* Age ≥18 years
* Histologically confirmed diagnosis of inoperable,locally advanced or metastatic cholangiocarcinoma (adenocarcinoma of intrahepatic,proximal extrahepatic,distal extrahepatic,gallbladder adenocarcinoma and periampullary bile duct adenocarcinoma).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Measurable disease criteria per RECIST v1.1.
* No prior chemotherapy or treatment with targeted therapy
* Formalin-fixed paraffin-embedded tumour and whole blood/plasma samples at diagnosis/study enrollment for biomarker studies.
* Adequate organ system function as specified in the protocol
* Female patients are allowed to participate provided they consent to avoid pregnancy throughout the course of the trial and 1 month after the last administration of the drug, if they are surgically sterilized or menopausal.

Exclusion Criteria:

* Prior malignancy.Subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma or indolent prostate cancer are eligible (even if they are receiving antihormonal therapy).
* Central nervous system (CNS) metastases at baseline, with the exception of those subjects who have previously-treated CNS metastases are asymptomatic and have no requirement for steroids or enzyme-inducing anticonvulsants in the past 6 months.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal, 28 days prior to study treatment initiation.
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including malabsorption syndrome, major resection of the stomach
* Corrected QT interval (QTc) >480 milliseconds using Bazett's formula
* History of myocardial infarction, unstable angina, symptomatic peripheral vascular disease or Class II,III or IV congestive heart failure, as defined by the New York Heart Association (NYHA) or cardiac angioplasty or stenting within the past 6 months
* Newly-diagnosed hypertension or history of poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 millimeters of mercury (mmHg)or diastolic blood pressure (DBP) of ≥90mmHg].
* History of cerebrovascular accident including transient ischemic attack(TIA),pulmonary embolism or untreated deep venous thrombosis(DVT) within the past 6 months.Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
* Major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture,or ulcer (procedures such as catheter placement not considered to be major).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage
* Recent hemoptysis (≥ ½ teaspoon of red blood within 8 weeks of first dose of study drug).
* Any serious and/or unstable pre-existing medical,psychiatric, or other condition that could interfere with subject's safety,provision of informed consent,or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug(whichever is longer) prior to the first dose of study drug and for the duration of the study
* Radiation therapy,surgery or tumor embolization within 14 days prior to the first dose of pazopanib
* Administration of any non-oncologic investigational study drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment.
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-06-28 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | At an average of 6 months for each patient
  Imaging evaluation for the determination of response to treatment will be performed every 8 weeks

SECONDARY OUTCOMES:
Evaluation of Progression-Free Survival (PFS) | PFS will be calculated from the date of treatment initiation to the date of disease progression or date of death, assessed up to 48 months
Evaluation of 6-month Progression-Free Survival rate (6-month PFS rate) | Assessed up to 6 months
  The aim is to determine the rate of PFS in patients, at 6 months of treatment
Evaluation of Overall Survival (OS) | OS will be calculated from the date of treatment initiation to the date of death from any cause, assessed up to 48 months.
Assessment of safety and tolerability | Assessed up to 48 months
  Distribution of Adverse Events (AEs) according to severity grade. Evaluation of AEs will be performed every 21 days (per treatment cycle) throughout the course of treatment
Evaluation of Quality of Life (QoL) | Assessed up to 9 months
  Quality of Life Questionnaires will be filled out before treatment initiation, every 8 weeks and at the end of treatment
Evaluation of potential prognostic and/or predictive biomarkers in tissue and blood samples | Tumor blocks and blood samples will be collected at baseline
  The following biomarkers will be analyzed:
  In bioptic material:
  * Stem Cell Factor (KIT)
  * Vascular Endothelial Growth Factor Receptor-2 (VEGF-2)
  * Vascular Endothelial Growth Factor Receptor-3 (VEGF-3)
  In peripheral blood/plasma:
  * Interleukin 8
  * Interleukin 12
  * Hepatocyte growth factor
  There may be additions to the biomarkers to be analyzed, dependent on the clinical and bibliographical data

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sgouros, MD, Study Chair — 3rd Dept of Medical Oncology, Agii Anargiri Cancer Hospital
Locations (17):
- Greece (17):
  - 2nd Dept of Internal Medicine, Agios Savvas Cancer Hospital, Athens
  - Dept of Medical Oncology, 251 General Air Force Hospital, Athens
  - 2nd Dept of Internal Medicine, General Hospital of Athens "Hippokratio", Athens
  - Oncology Dept, 2nd Surgyc Clinic, Aretaieio Hospital, Athens
  - Oncology Section, Dept of Clinical Therapeutics, General Hospital of Athens "Alexandra", Athens
  - Division of Oncology, 2nd Dept of Internal Medicine, Propaedeutic, University Hospital "Attikon", Athens
  - 2nd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens
  - 3rd Dept of Medical Oncology, Agii Anargiri Cancer Hospital, Athens
  - 3rd Dept of Medical Oncology, Hygeia Hospital, Athens
  - 1st Dept of Medical Oncology, Metropolitan Hospital, Athens
  - 2nd Dept of Medical Oncology, Metropolitan Hospital, Athens
  - Dept of Medical Oncology, University Hospital of Heraklion, Heraklion
  - Dept of Medical Oncology, Ioannina University Hospital, Ioannina
  - Division of Oncology, Dept of Internal Medicine, University Hospital of Patras, Pátrai
  - 2nd Dept of Medical Oncology, EUROMEDICA General Clinic of Thessaloniki, Thessaloniki
  - Dept of Medical Oncology, Papageorgiou General Hospital, Thessaloniki
  - Dept of Medical Oncology, Thermi Clinic S.A, Thessaloniki